CLINICAL TRIAL: NCT05168709
Title: A Single-arm Clinical Trial to Investigate COVID-19 Specific Vaccine and Heterologous Immunity in the Melbourne Infant Study of BCG for Allergy and Infection Reduction (COSI BAIR)
Brief Title: Investigating COVID-19 Vaccine Immunity in Children in the Melbourne Infant Study of BCG for Allergy and Infection Reduction
Acronym: COSI BAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 81771
Record Dates: First submitted 2021-12-22; First posted 2021-12-23 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Vaccine Reaction; Immunization; Infection
Keywords: Non-specific effects; COVID-19 vaccination; paediatric vaccination; heterologous immunity; mRNA vaccine
MeSH Terms: conditions — COVID-19; Infections | interventions — BNT162 Vaccine; RNA, Messenger

STUDY DESIGN:
Intervention Model Description: This trial is a non-controlled single-arm post-marketing exploratory trial where the approved COVID-19 vaccine will be used to determine whether COVID-19 vaccination alters heterologous (non-COVID-19-specific) immunity in children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Approved COVID-19 vaccination (Experimental): The approved COVID-19 vaccination arm will receive the COMIRNATY™ (tozinameran - BNT162b2 [mRNA]) COVID-19 VACCINE. The dose, strength of the dose unit, dosing interval and dosing period of tozinameran used in this trial will be as approved by the Therapeutic Goods Administration (TGA) and recommended by the Australian Technical Advisory Group on Immunisation (ATAGI) for children aged 5 to <12 years of age. The recommended dose of tozinameran for this age group is 10 µg (0.2 mL) and the recommended schedule is 2 doses, 8 weeks apart. Therefore two tozinameran doses of 10µg (0.2 mL) will be administered intramuscularly 8-weeks apart as part of this arm of the trial.
  Interventions: Biological: Tozinameran

INTERVENTIONS:
Biological: Tozinameran — Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cell-free in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
  Other Names: COMIRNATY; BNT162b2 [mRNA]; Pfizer COVID-19 Vaccine

SUMMARY:
The COSI BAIR trial will involve approximately 60 children, aged 5 to 8 years old, comprising a subset of participants from the Melbourne Infant Study BCG for Allergy and Infection Reduction (MIS BAIR) randomised controlled trial. The overall aim of this trial is to investigate the specific and heterologous effects of COVID-19 vaccination on immunity in children. COSI BAIR will aim to recruit its participants from the MIS BAIR Bacillus Calmette-Guérin (BCG)-naïve group. These children will be followed up until 28 days after their final Coronavirus Disease 2019 (COVID-19) vaccination.

Venous blood samples will be collected at two study visits, at Murdoch Children's Research Institute (MCRI):

1. Day 0 - baseline (day of COVID-19 vaccination #1), and
2. Day 84 (28 days after COVID-19 vaccination #2).

ELIGIBILITY:
Inclusion Criteria:

* Age between five and eleven years (i.e. prior to the twelfth birthday) at the time of enrolment,
* Participant who was randomised in the MIS BAIR trial, and

  * Was randomly allocated to receive and received BCG as part of the MIS BAIR trial, OR,
  * Was randomly allocated to not receive and did not receive BCG;
* Is an individual whose parent/legally acceptable representative (LAR) consented to be contacted about future ethically approved research, during the MIS BAIR trial consent process, AND
* Has a parent/LAR capable of understanding the parent/LAR information statement and consent form (PICF) document and providing consent on the participant's behalf.

Exclusion Criteria:

* Has a known hypersensitivity to the active ingredient or any of the excipients in tozinameran,
* Has a prior polymerase chain reaction (PCR)-confirmed diagnosis of COVID-19 whether symptomatic or not,
* Has received a COVID-19 vaccine (approved by the TGA or otherwise) prior to trial enrolment,
* An individual and/or parent/legally acceptable representative who is unwilling or unable to give written informed consent,
* An individual and/or parent/legally acceptable representative who is unwilling or unable to consent to attend all scheduled study visits,
* An individual and/or parent/LAR who is unwilling or unable to give consent for blood samples to be taken from the trial participant at each study visit, and
* Has or has had a clinically significant medical morbidity (e.g. immunocompromised because of congenital or acquired disorders or immunosuppressive medical treatment; a bleeding disorder; a recent history of inflammatory cardiac illness within the past 6 months, e.g., myocarditis, pericarditis, endocarditis, acute rheumatic fever (with active myocardial inflammation) or acute rheumatic heart disease, or acute decompensated heart failure), and
* Has received BCG at any other time than as part of the MIS BAIR trial.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline of in vitro whole blood stimulation cytokine responses to COVID-19 specific and heterologous stimulants | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  The difference in cytokine concentrations between those measured on the day of first vaccination and 28 days after second vaccination is the primary outcome measure

SECONDARY OUTCOMES:
Mean change from baseline of anti-SARS-CoV-2 antibody titres | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  The difference in anti-SARS-CoV-2 antibody titres between those measured on the day of first vaccination and 28 days after second vaccination is outcome measure 2
Mean change from baseline of SARS-CoV-2-reactive T cell responses | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  The difference in SARS-CoV-2-reactive T cell responses, as measured by interferon-gamma producing units, between those measured on the day of first vaccination and 28 days after second vaccination is outcome measure 3
Correlation of serological profiling of previous viral infections and antiviral responses, and post-vaccination anti-SARS-CoV-2 antibody titres | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  Pearson product-moment correlation coefficient of all trial participants' serological profiling of previous viral infections and antiviral responses on the day of first COVID-19 vaccination and anti-SARS-CoV-2 antibody titres measured at 28 days after second vaccination is outcome measure 4. Previous viral infection organisms considered will include SARS-CoV-1, Middle East Respiratory Syndrome Coronavirus and circulating coronaviruses (eg. human coronavirus HKU1).
Correlation of serological profiling of vaccine-preventable disease antibody responses and post-vaccination anti-SARS-CoV-2 antibody titres | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  Pearson product-moment correlation coefficient of all trial participants' vaccine-preventable disease antibody responses on the day of first COVID-19 vaccination and anti-SARS-CoV-2 antibody titres measured at 28 days after second vaccination is outcome measure 5. Vaccine-preventable disease organisms examined will include Haemophilus influenzae B, Streptococcus pneumoniae and measles.
Correlation of whole blood cytokine responses to vaccine-preventable disease antigens and post-vaccination anti-SARS-CoV-2 antibody titres | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  Pearson product-moment correlation coefficient of all trial participants' whole blood cytokine responses to vaccine-preventable disease antigens on the day of first COVID-19 vaccination and anti-SARS-CoV-2 antibody titres measured at 28 days after second vaccination is outcome measure 6. Vaccine-preventable disease organisms examined will include Haemophilus influenzae B, Streptococcus pneumoniae and measles.
Mean change from baseline of vaccine-preventable disease antibody titres | Day 0 (the day of the first COVID-19 vaccine dose) to day 84 (28 days after the second COVID-19 vaccine dose)
  The difference in vaccine-preventable disease antibody titres between those measured on the day of first vaccination and 28 days after second vaccination is outcome measure 7. Vaccine-preventable disease organisms examined will include Haemophilus influenzae B, Streptococcus pneumoniae and measles.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Curtis, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Melbourne Children's campus, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
At the time of article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access:
  * Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures and appendices), and
  * Trial protocol, PICF, analytic code
  We may share the information and samples we collect with other researchers within Australia and/or overseas to increase our understanding of COVID-19 and COVID-19 vaccination and other infections. The location of data/samples sent overseas is not yet determined. Data and samples would be sent identifiable only by a study number so that the child's identity is not disclosed to these researchers. Any data or samples sent to researchers outside of Australia will not be covered by Australian regulations.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Following the completion and analysis of the trial, the data will be retained long-term following the mandatory archive period for use in future research projects. The retention period will be for at least 15 years post-trial completion or until the child is aged 25 years (whichever is later). The Sponsor-Investigator and/or delegate will be the custodians during the archive period. Following the end of the archival period, the data will be disposed of.
Access Criteria: * Must pertain to ethically approved research
  * Must be from a recognised institution
  * Must be willing to share the aims, outcomes and outcomes measures of the secondary analyses
  * Must ask for consent from the COSI BAIR principal investigators
  * Must be approved by the COSI BAIR Sponsor-Investigator

REFERENCES:
- [Background] Freyne B, Messina NL, Donath S, Germano S, Bonnici R, Gardiner K, Casalaz D, Robins-Browne RM, Netea MG, Flanagan KL, Kollmann T, Curtis N; Melbourne Infant Study: BCG for Allergy and Infection Reduction (MIS BAIR) Group. Neonatal BCG Vaccination Reduces Interferon-gamma Responsiveness to Heterologous Pathogens in Infants From a Randomized Controlled Trial. J Infect Dis. 2020 Jun 11;221(12):1999-2009. doi: 10.1093/infdis/jiaa030. PMID 31990350
- [Background] Freyne B, Donath S, Germano S, Gardiner K, Casalaz D, Robins-Browne RM, Amenyogbe N, Messina NL, Netea MG, Flanagan KL, Kollmann T, Curtis N. Neonatal BCG Vaccination Influences Cytokine Responses to Toll-like Receptor Ligands and Heterologous Antigens. J Infect Dis. 2018 May 5;217(11):1798-1808. doi: 10.1093/infdis/jiy069. PMID 29415180
- [Background] Messina NL, Pittet LF, Gardiner K, Freyne B, Francis KL, Zufferey C, Abruzzo V, Morrison C, Allen KJ, Flanagan KL, Ponsonby AL, Robins-Browne R, Shann F, South M, Vuillermin P, Donath S, Casalaz D, Curtis N. Neonatal Bacille Calmette-Guerin Vaccination and Infections in the First Year of Life: The MIS BAIR Randomized Controlled Trial. J Infect Dis. 2021 Oct 13;224(7):1115-1127. doi: 10.1093/infdis/jiab306. PMID 34146093
- [Background] Messina NL, Gardiner K, Donath S, Flanagan K, Ponsonby AL, Shann F, Robins-Browne R, Freyne B, Abruzzo V, Morison C, Cox L, Germano S, Zufferey C, Zimmermann P, Allen KJ, Vuillermin P, South M, Casalaz D, Curtis N. Study protocol for the Melbourne Infant Study: BCG for Allergy and Infection Reduction (MIS BAIR), a randomised controlled trial to determine the non-specific effects of neonatal BCG vaccination in a low-mortality setting. BMJ Open. 2019 Dec 15;9(12):e032844. doi: 10.1136/bmjopen-2019-032844. PMID 31843845
- [Background] Zimmermann P, Donath S, Perrett KP, Messina NL, Ritz N, Netea MG, Flanagan KL, van der Klis FRM, Curtis N; MIS BAIR group. The influence of neonatal Bacille Calmette-Guerin (BCG) immunisation on heterologous vaccine responses in infants. Vaccine. 2019 Jun 19;37(28):3735-3744. doi: 10.1016/j.vaccine.2019.03.016. Epub 2019 May 29. PMID 31153688
- [Background] Pittet LF, Messina NL, Gardiner K, Freyne B, Abruzzo V, Francis KL, Morrison C, Zufferey C, Vuillermin P, Allen KJ, Ponsonby AL, Robins-Browne R, Shann F, Flanagan KL, Phillips R, Donath S, Casalaz D, Curtis N. Prevention of infant eczema by neonatal Bacillus Calmette-Guerin vaccination: The MIS BAIR randomized controlled trial. Allergy. 2022 Mar;77(3):956-965. doi: 10.1111/all.15022. Epub 2021 Aug 9. PMID 34309859
- See also: MIS BAIR trial website. Participants for COSI BAIR will be recruited from this trial population. — https://www.mcri.edu.au/misbair